CLINICAL TRIAL: NCT00567801
Title: Prospektive, Randomisierte Multicenter-Studie Zur Optimierung Der Therapie Der Akuten Ischämie Der Unteren Extremitäten Durch Die Kontrollierte Extremitätenreperfusion (Prospective, Randomized Multicenter - Study for Optimization of Therapy of the Acute Ischemic Limb by Controlled Reperfusion)
Brief Title: CRAIL - Controlled Reperfusion of the Acutely Ischemic Limb
Acronym: CRAIL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Collaborators: Dr. Köhler Chemie (Alsbach-Hähnlein, Germany) (Unknown); HP-Medica (Augsburg, Germany) (Unknown); GEA (Frederiksberg, Denmark) (Unknown); Kardialagut (München, Germany) (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S 991228
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2008-07-28 (Estimated); Status verified 2008-07

CONDITIONS: Lower Extremity Ischemia
Keywords: Lower Extremity; Ischemia
MeSH Terms: conditions — Ischemia | interventions — Thrombectomy; Embolectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): conventional embolectomy/thrombectomy
  Interventions: Procedure: conventional embolectomy/thrombectomy
- 2 (Experimental): embolectomy/thrombectomy with controlled reperfusion
  Interventions: Procedure: embolectomy/thrombectomy with controlled reperfusion

INTERVENTIONS:
Procedure: conventional embolectomy/thrombectomy
  Arms: 1
Procedure: embolectomy/thrombectomy with controlled reperfusion
  Arms: 2

SUMMARY:
The purpose of this study is to prove the findings of a preliminary study which strongly suggest the hypothesis that the result of conventional embolectomy for acute, severe lower-limb ischemia can be improved by controlled reperfusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Patients with arterial occlusion of one or both lower limbs with acute decompensated ischemia (Rutherford IIA to III)
* Informed consent of the patient

Exclusion Criteria:

* Previous attempt of recanalisation (e.g. lysis therapy)
* Known A. poplitea aneurysm of the affected extremity
* Severe heart failure NYHA IV
* Known atrial thrombus
* Terminal renal insufficiency (creatinine >10mg/dl or current dialysis therapy, previous transplantation of kidney)
* Hypersensitivity to allopurinol
* Hypersensitivity to one component part of the reperfusion solution
* Participation in a clinical trial during the study or 30 days before
* Pregnancy or lactation
* Patient incapable of contracting or not able to understand the character, meaning and consequences of the clinical trial
* Abuse to drugs or alcohol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2002-09; Primary Completion 2009-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Amputation-free survival | 28 days

SECONDARY OUTCOMES:
Neurological status (motor function, sensor function) of ischemic limb | 4 weeks
Systemic complications in both therapy groups | 4 weeks
Tolerance of reperfusion solution | 4 weeks
Lethality | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Friedhelm Beyersdorf, Prof. Dr., Principal Investigator — Department of Cardiovascular Surgery, University Medical Center Freiburg
Locations (23):
- Austria (2):
  - Universität Innsbruck, Innsbruck
  - St. Johanns-Spital Salzburg, Salzburg
- Germany (21):
  - University Medical Center Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Städtisches Klinikum Karlsruhe, Karlsruhe, Baden-Wurttemberg
  - Klinikum Lahr, Lahr, Baden-Wurttemberg
  - Klinikum Villingen-Schwenningen, Villingen-Schwenningen, Baden-Wurttemberg
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Universitätsklinikum Bonn, Bonn
  - Kreisklinikum Donaueschingen, Donaueschingen
  - St. Johannes-Hospital Dortmund, Dortmund
  - Marienhospital Altenessen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - St. Marien-Hospital Buer, Gelsenkirchen, Gelsenkirchen
  - Universitätsklinikum Giessen, Giessen
  - Herzzentrum Göttingen, Göttingen
  - Uniklinik Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Kiel, Kiel
  - Park-Krankenhaus Leipzig, Leipzig
  - Universitätsklinikum Lübeck, Lübeck
  - Universitätsklinikum Mainz, Mainz
  - Klinikum E. v. Bergmann Potsdam, Potsdam
  - Universitätsklinikum Rostock, Rostock
  - Hegau-Klinikum Singen, Singen

REFERENCES:
- [Background] Wilhelm MP, Schlensak C, Hoh A, Knipping L, Mangold G, Dallmeier Rojas D, Beyersdorf F. Controlled reperfusion using a simplified perfusion system preserves function after acute and persistent limb ischemia: a preliminary study. J Vasc Surg. 2005 Oct;42(4):690-4. doi: 10.1016/j.jvs.2005.05.055. PMID 16242556